CLINICAL TRIAL: NCT03229642
Title: The Effects of Repetitive Transcranial Magnetic Stimulation in Patients With Opioid Use Disorders: Analysis of Clinical Outcomes, Functional Magnetic Resonance Imaging, Biomarkers, and Neuropsychological Tests
Brief Title: Repetitive Transcranial Magnetic Stimulation in Patients With Opioid Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Tzu-Yun Wang, Doctor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-BR-105-094
Record Dates: First submitted 2017-07-11; First posted 2017-07-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Transcranial Magnetic Stimulation; Heroin Dependence
Keywords: repetitive transcranial magnetic stimulation; opioid use disorder; craving; functional magnetic resonance imaging; neuropsychological tests
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS treatment (Experimental): The rTMS parameters were as follows: 15Hz frequency, pulse intensity 100% of the rMT, 60 pulses per train, inter train pause of 26 sec, 40 stimulation trains, and 2400 total pulses for a total duration of 20 min. The patients received one rTMS session per day during the first five days of treatment, and then twice a week for the following three weeks, for a total of 11 rTMS sessions.
  Interventions: Device: Active rTMS
- Sham rTMS treatment (Sham Comparator): The rTMS parameters were as follows: 15Hz frequency, pulse intensity 100% of the rMT, 60 pulses per train, inter train pause of 26 sec, 40 stimulation trains, and 2400 total pulses for a total duration of 20 min, with a figure-of-eight sham coil. The patients received one rTMS session per day during the first five days of treatment, and then twice a week for the following three weeks, for a total of 11 rTMS sessions.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — The stimulator device was a Magstim super rapid magnetic stimulator (Magstim Company, Ltd., Wales, United Kingdom) with 4 booster modules equipped with a 70-mm air-cooled figure-eight-shaped coil. We performed rTMS on the left dorsolateral prefrontal cortex (DLPFC).The TMS parameters were as follows: 15Hz frequency, pulse intensity 100% of the rMT, 60 pulses per train, inter train pause of 26 sec, 40 stimulation trains, and 2400 total pulses for a total duration of 20 min. The patients received one rTMS session per day during the first five days of treatment, and then twice a week for the following three weeks, for a total of 11 rTMS sessions. The sham group was administered rTMS with the same parameters, but using a figure-of-eight sham coil.
  Arms: Active rTMS treatment
Device: Sham rTMS — The stimulator device was a Magstim super rapid magnetic stimulator (Magstim Company, Ltd., Wales, United Kingdom) with 4 booster modules equipped with a 70-mm air-cooled figure-eight-shaped coil. We performed rTMS on the left dorsolateral prefrontal cortex (DLPFC).The TMS parameters were as follows: 15Hz frequency, pulse intensity 100% of the rMT, 60 pulses per train, inter train pause of 26 sec, 40 stimulation trains, and 2400 total pulses for a total duration of 20 min. The patients received one rTMS session per day during the first five days of treatment, and then twice a week for the following three weeks, for a total of 11 rTMS sessions. The sham group was administered rTMS with the same parameters, but using a figure-of-eight sham coil.
  Arms: Sham rTMS treatment

SUMMARY:
Opioid use disorder (OUD) is prevalent and causes substantial health and social burdens. Although evidence have showed the effectiveness of opioid agonist maintenance therapy in OUD, high drop-out rate and the requirement of continuing use of opioid agonists are the major problems. Therefore, to develop novel treatment for OUD is important.

Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive method of brain stimulation used to treat a variety of neuropsychiatric disorders. Recent studies showed that there may be potential therapeutic effects in rTMS for addictive disorder, including reducing craving and substance use severity. The underlying mechanisms of rTMS in treating addictions may involve increased dopamine function in corticomesolimbic brain circuits and modulation of neural activity in brain circuits that relevant to addiction. However, the treatment results of rTMS in OUD were lacked, and the analysis in functional brain imaging study, neuropsychological tests and other potential biomarkers under rTMS treatment were limited, too.

Thus, the investigators will conduct the add-on double-blinded, sham-controlled study rTMS treatment in 40-60 patients with OUD under methadone maintenance therapy. Patients will be allocated to active and sham rTMS in a 1 : 1 ratio, and participants will receive rTMS on the left dorsolateral prefrontal cortex (DLPFC) (15 Hz frequency, 4 seconds per train, inter-train interval of 26 seconds, 40 trains per session, total 11 sessions in 4 weeks). The treatment response, urine drug tests, craving scales and side effects to evaluate the therapeutic effects of rTMS will be examined. Neuropsychological assessments, functional magnetic resonance imaging (fMRI) and tests for potential biomarkers of immune parameters will also be measured during 12-weeks follow up. The study results will provide the important data in whether rTMS add-on methadone maintenance therapy is able to 1) reduce heroin use; 2) reduce craving for heroin; 3) be an effective treatment for OUD, and 4) be associated with improvement in fMRI, biological markers and psychological tests.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient or legal representative.
2. Male or female patient aged ≧20 and ≦65 years.
3. A diagnosis of OUD according to DSM criteria made by a specialist in psychiatry.
4. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

1. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study.
2. Females who are pregnant or lactation.
3. Current evidence of an uncontrolled and/or clinically significant medical condition, e.g.,cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation.
4. History of seizure or epilepsy.
5. History of neurological diseases or traumatic brain injury.
6. Suicidal attempts or risks during screen or study period.
7. Presence of devices, e.g. pace-makers, cochlear prosthesis, neuro-stimulators, magnetic cochlear prosthesis, intraocular metallic fragments.
8. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to the first intervention of the double-blinded treatment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The treatment retention rate | 12 weeks
  To compare the treatment retention rate between the active and sham rTMS groups from baseline to endpoint (12 weeks).
The treatment attendance rate | 12 weeks
  To compare the treatment attendance rate between the active and sham rTMS groups from baseline to endpoint (12 weeks).
Urinary assessment | 12 weeks
  Urinary morphine examinations will be measured at every visit. The rate of positive urinary morphine tests will be compared between active and sham rTMS groups in 12 weeks of follow up.

SECONDARY OUTCOMES:
fMRI | 5 weeks
  The fMRI scan will be done at initial screen and at week 5 (after rTMS treatment) with resting-state fMRI and task activation fMRI with an IGT.
Immunological markers | 12 weeks
  Twenty milliliters of blood will be drawn from each participant. Plasma will be isolated from the whole blood after it has been centrifuged at 3000 g for 15 min at 4℃, and the will be immediately stored at -80℃. Cytokine and BDNF levels will be quantified using an antibody pair assay system (Flexia; BioSource Intl., Camarillo, CA). Sample processing and data analysis will be done according to the manufacturer's instructions.
  The immunological parameters that we intend to analyze will include TNF-α, CRP, TGF-β1, IL-8, Il-10 and BDNF. The immunological markers will be measured from baseline to endpoint (week 12) in each patient group.
Wechsler Memory Scale - third edition(WMS-III) | 12 weeks
  WMS-III will be tested at initial screen and at the end of study (week 12) and compared between the active and sham rTMS groups.
Wisconsin Card Sorting Test(WCST) | 12 weeks
  WCST will be tested at initial screen and at the end of study (week 12) and compared between the active and sham rTMS groups.
Continuous performance tests(CPT) | 12 weeks
  CPT will be tested at initial screen and at the end of study (week 12) and compared between the active and sham rTMS groups.
Side effect checklist | 12 weeks
  To compare the side effect profiles using side effect checklist between the active and sham rTMS groups from baseline to endpoint (12 weeks).
Assessment of craving | 12 weeks
  To compare the severity of craving between the active and sham rTMS groups from baseline to endpoint (12 weeks).
17-item Hamilton Depression Rating Scale (HDRS) | 12 weeks
  To compare the mood symptoms between the active and sham rTMS groups from baseline to endpoint (12 weeks).
World Health Organization's Quality of Life Assessment-Brief of Taiwan (WHOQOL-BREF TW) | 12 weeks
  To compare the life quality (using WHOQOL-BREF TW) between the active and sham rTMS groups from baseline to endpoint (12 weeks).
Family APGAR index | 12 weeks
  To compare the level of family support (using family APGAR index) between the active and sham rTMS groups from baseline to endpoint (12 weeks).
The Opiate Treatment Index (OTI) | 12 weeks
  To compare the OTI tween the active and sham rTMS groups from baseline to endpoint (12 weeks).
Clinical Global Impressions (CGI) | 12 weeks
  To compare the CGI tween the active and sham rTMS groups from baseline to endpoint (12 weeks).
Barratt Impulsiveness Scale(BIS) | 12 weeks
  To compare the BIS tween the active and sham rTMS groups from baseline to endpoint (12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yun Wang, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Tsai TY, Wang TY, Liu YC, Lee PW, Chang WH, Lu TH, Tseng HH, Lee SY, Chang YH, Yang Y, Chen PS, Chen KC, Yang YK, Lu RB. Add-on repetitive transcranial magnetic stimulation in patients with opioid use disorder undergoing methadone maintenance therapy. Am J Drug Alcohol Abuse. 2021 May 4;47(3):330-343. doi: 10.1080/00952990.2020.1849247. Epub 2021 Jan 10. PMID 33426970